CLINICAL TRIAL: NCT05687890
Title: A Randomized, Double Blind, Placebo Parallel Controlled, 2 Cohorts, Multicenter Phase II Study to Investigate the Safety and Efficacy of SC0062 Capsule in Patients With Chronic Kidney Disease With Albuminuria
Brief Title: A Study to Evaluate the Efficacy and Safety of SC0062 in the Treatment of Chronic Kidney Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biocity Biopharmaceutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SC0062-202
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Kidney Disease; IgA Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies; Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SC0062 low dose group (Experimental): Subjects will take two capsules daily for 24 weeks during the treatment period
  Interventions: Drug: SC0062 low dose
- SC0062 medium dose group (Experimental): Subjects will take two capsules daily for 24 weeks during the treatment period
  Interventions: Drug: Placebo of SC0062; Drug: SC0062 medium dose
- SC0062 high dose group (Experimental): Subjects will take two capsules daily for 24 weeks during the treatment period
  Interventions: Drug: SC0062 high dose
- Placebo of SC0062 group (Placebo Comparator): Subjects will take two capsules daily for 24 weeks during the treatment period
  Interventions: Drug: Placebo of SC0062

INTERVENTIONS:
Drug: Placebo of SC0062 — Subjects will take two capsules daily of one of those which are SC0062 low dose, SC0062 medium dose, SC0062 high dose or placebo for 24 weeks during the treatment period
  Arms: Placebo of SC0062 group; SC0062 medium dose group
Drug: SC0062 low dose — Subjects will take two capsules daily of one of those which are SC0062 low dose, SC0062 medium dose, SC0062 high dose or placebo for 24 weeks during the treatment period
  Arms: SC0062 low dose group
Drug: SC0062 medium dose — Subjects will take two capsules daily of one of those which are SC0062 low dose, SC0062 medium dose, SC0062 high dose or placebo for 24 weeks during the treatment period
  Arms: SC0062 medium dose group
Drug: SC0062 high dose — Subjects will take two capsules daily of one of those which are SC0062 low dose, SC0062 medium dose, SC0062 high dose or placebo for 24 weeks during the treatment period
  Arms: SC0062 high dose group

SUMMARY:
This is a phase II study to investigate the safety, preliminary efficacy and pharmacokinetics of SC0062 capsule in patients with chronic kidney disease (diabetic kidney disease and IgA nephropathy)with albuminuria compared to matching placebo.

DETAILED DESCRIPTION:
This multicenter, randomized, double blind, placebo parallel controlled, 2 cohorts phase II study will contain 2 cohorts:

Cohort 1: diabetic kidney disease

Cohort 2: biopsy-proven IgAN

In each cohort, approximately 120 patients will be randomized to receive SC0062 or placebo daily for 24 weeks.

The objective of this study is to evaluate the preliminary efficacy and safety of SC0062 capsules compared to placebo in patients with chronic kidney disease (diabetic kidney disease and IgA nephropathy) with albuminuria who are treated with the maximum tolerated labeled dose renin-angiotensin system inhibitor (RASi).

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent voluntarily, and fully understand and comply with the relevant procedures of the test;
2. Age of ≥ 18 years old, gender is not limited;
3. Patients with chronic kidney disease (CKD) stage G1~G3 with albuminuria, requirements:

   1. eGFR ≥ 30 mL/min/1.73m^2 at Screening based on the CKD-EPI equation (2009).
   2. RAS inhibitor therapy (ACEi and/or ARB) has been administered for at least 12 weeks and the maximally tolerated dose has been stable for at least 4 weeks prior to randomization; If an SGLT2i is prescribed, the dose must be stable for at least 8 weeks prior to randomization.
   3. Cohort 1: Diagnosed with type 2 diabetes mellitus and receiving at least one hypoglycemic agent in the 12 months prior to randomization; In accordance with the diagnostic criteria of DKD, urine albumin to creatinine ratio (UACR) ≥300 mg/g before randomization.
   4. Cohort 2: Biopsy-proven IgA nephropathy; Urine protein-creatinine ratio (UPCR) ≥0.75 g/g or urine protein excretion rate ≥ 1.0 g/24h before randomization.
4. Laboratory parameters meet the following criteria:

   1. Serum albumin ≥30 g/L;
   2. Hemoglobin value ≥90 g/L; Platelet ≥80×10^9/L;
   3. Brain natriuretic peptide (BNP) ≤ 200 pg/mL or N-terminal pro-B-type natriuretic peptide (NT-proBNP) ≤ 600 pg/mL;
   4. Blood potassium ≤ 5.5 mmol/L;
   5. Systolic blood pressure (SBP) ≤140 mmHg; Diastolic blood pressure (DBP) ≤90 mmHg;
   6. Hemoglobin A1c (HbA1c) ≤ 10% (cohort 1)/Hemoglobin A1c (HbA1c) < 6.5% (cohort 2);
   7. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2×ULN; Total bilirubin ≤1.5ULN;
5. All participants should follow protocol defined contraceptives procedures.

Exclusion Criteria:

1. Women who were pregnant or breastfeeding; A WOCBP who has a positive blood pregnancy test prior to randomization;
2. Patients who are allergic to or are allergic to any component of the study drug (SC0062 capsules);
3. Systemic use of corticosteroids or immunosuppressants for more than 2 weeks within 3 months prior to randomization; with exceptions as follows: Topical or intra-articular, intranasal, and inhaled glucocorticoids; on stable doses of hydroxychloroquine for at least 8 weeks.
4. Type 1 diabetes or other specific types of diabetes;
5. Secondary IgA nephropathy;
6. Clinical suspicion of rapidly progressive glomerulonephritis (RPGN);
7. Diagnosed with nephrotic syndrome;
8. Have a history of pulmonary hypertension (WHO Group 1), idiopathic pulmonary fibrosis or any lung disease requiring oxygen therapy (e.g., chronic obstructive pulmonary disease, emphysema, pulmonary edema, etc.);
9. Subjects who had received endothelin receptor antagonist in the past;
10. History of moderate or severe edema, non-traumatic facial edema, or myxoid edema within the 6 months prior to randomization;
11. History of orthostatic hypotension within 6 months prior to randomization;
12. History of clinically significant cirrhosis;
13. History of heart failure NYHA Class III~IV; exacerbation heart failure or acute coronary syndrome within 6 months prior to randomization;
14. History of renal transplantation or other organ transplantation;
15. Hypothyroidism (except subclinical hypothyroidism or stable hypothyroidism after hormone replacement therapy);
16. Patients who have the potential to interfere with oral drug absorption, such as subtotal gastrectomy, clinically severe gastrointestinal disease, or certain types of bariatric surgery, such as gastric bypass surgery, that do not involve simply separating the stomach into a separate chamber, such as gastric banding surgery;
17. Use of potent CYP3A4 inducers (e.g., rifampicin, carbamazepine, phenytoin, phenobarbital, St. John's Burt) and potent CYP3A4 inhibitors (e.g., itraconazole, ketoconazole, voriconazole, clarithromycin, telomycin, nefazodone, ritonavir, saquinavir) within 1 month before randomization;
18. Active hepatitis B; active hepatitis C; active syphilis; positive HIV serum reaction.
19. Malignancy within the past 5 years (Except for treated basal cell carcinoma of the skin, effectively resected squamous cell carcinoma of the skin, colon polyps, or cervical cancer in situ that do not require ongoing treatment);
20. Alcohol or drug abuse or dependence, or a history of psychological disorder;
21. Participants participated in clinical trials of other investigational drugs or medical devices within 3 months prior to randomization;
22. Any other clinically significant clinical condition, or medical history may interfere with the subject's safety, study evaluation, and/or study procedures per the judgment by the investigator;
23. The investigator believes that the subject has any other reasons for not being eligible to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in urine albumin creatinine ratio (UACR) | Week 12
  Change from baseline at Week 12 in urine albumin creatinine ratio (UACR) in Cohort 1
Changes in urine protein creatinine ratio (UPCR) | Week 12
  Change from baseline at Week 12 in urine protein creatinine ratio (UPCR) in Cohort 2

SECONDARY OUTCOMES:
Change in urine albumin creatinine ratio (UACR) by visit | Week 2, week 4, week 8, week 12, week 16, week 20, week 24
  Change in urine albumin creatinine ratio (UACR) after treatment
Change in urine protein creatinine ratio (UPCR) by visit | Week 2, week 4, week 8, week 12, week 16, week 20, week 24
  Change in urine protein creatinine ratio (UPCR) after treatment
Changes in glomerular filtration rate (eGFR) | Week 2, week 4, week 8, week 12, week 16, week 20, week 24
  Change in glomerular filtration rate (eGFR) from baseline to end of study
Change of 24-hour urine albumin excretion rate (UAER) | Week 12, week 24
  Change of 24-hour urine albumin excretion rate (UAER) at Week 12 and Week 24 in Cohort 1
Change of 24-hour urine protein excretion rate (UPER) | Week 12, week 24
  Change of 24-hour urine protein excretion rate (UPER) at Week 12 and Week 24 in Cohort 2
Percentage of subjects achieving UACR ≥30%, ≥40%, and ≥50% reduction from baseline | Week 12, week 24
  Percentage of subjects achieving UACR ≥30%, ≥40%, and ≥50% reduction at Week 12 and Week 24 in Cohort 1
Percentage of subjects achieving UPCR ≥30%, ≥40%, and ≥50% reduction from baseline | Week 12, week 24
  Percentage of subjects achieving UPCR ≥30%, ≥40%, and ≥50% reduction at Week 12 and Week 24 in Cohort 2

CONTACTS AND LOCATIONS:
Overall Officials: Jianghua Chen, Prof, Principal Investigator — Zhejiang University
Locations (1):
- 79 Qingchun Rd.,Shangcheng District, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Heerspink HJL, Du X, Xu Y, Zhang Y, Liu B, Bi G, Xu C, Luo Q, Wu H, Wan J, Cao L, Wang R, Fan Q, Cheng H, Xu L, Huang J, Zhong A, Peng Q, Hei Y, Wang Y, Zhou B, Zhang L, Chen J. The Selective Endothelin Receptor Antagonist SC0062 in IgA Nephropathy: A Randomized Double-Blind Placebo-Controlled Clinical Trial. J Am Soc Nephrol. 2025 Apr 1;36(4):657-667. doi: 10.1681/ASN.0000000538. Epub 2024 Oct 26. PMID 39462310
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639